CLINICAL TRIAL: NCT03926429
Title: A Bicentre Retrospective Study of Features and Outcomes of Patients With Reactive Arthritis
Brief Title: Features and Outcomes of Patients With Reactive Arthritis
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: FOPRA
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with reactive arthritis
  Interventions: Other: Standardised data collection

INTERVENTIONS:
Other: Standardised data collection — The following variables will be retrospectively assessed by medical record review using a standardised data collection form:demographics; gender, age; family or personal history of spondyloarthritis, psoriasis, uveitis, inflammatory bowel disease; clinical presentation; mono, oligo or polyarthritis, dactylitis, inflammatory joint pain, enthesopathy, axial symptoms, fever, extra-articular manifestations (conjunctivitis, anterior uveitis, circinate balanitis, skin rash); time interval between infection and musculoskeletal manifestations; causal microorganism if known, or triggering event; HLA-B27; radiographic sacroiliitis; treatments and outcomes (complete recovery at one year follow-up, relapse within 6 months after onset, or spondyloarthritis according to the ASAS criteria).

SUMMARY:
The aim of this study is to assess the incidence and the clinical and therapeutic characteristics of reactive arthritis and to compare them with those of a historical cohort. We hypothesised that improved hygiene together with prevention and treatment of sexually transmitted infections may have decreased the incidence of reactive arthritis.

ELIGIBILITY:
Inclusion Criteria:

* reactive arthritis diagnosed in one of the two rheumatology departments from Centre Hospitalier Lyon Sud or Besançon

Exclusion Criteria:

* presence of other known causes of arthritis, such as other defined spondyloarthritides, septic arthritis, Lyme disease, microcrystalline arthritis or rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active reactive arthritis
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of reactive arthritis in patients hospitalised in the rheumatology department | December 2014
  Incidence of reactive arthritis in patients hospitalised in the rheumatology department

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne COURY-LUCAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite